CLINICAL TRIAL: NCT05529264
Title: Human Intracranial Electrophysiology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Krzysztof Bujarski, Section Chief, Neurology, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY02001606
Record Dates: First submitted 2022-08-22; First posted 2022-09-07 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Invasive EEG (electrodes are implanted in a participant's brain) (Experimental): Patients with intracranial electrodes (electrodes are implanted in a participant's brain) undergoing pre-surgical evaluation for clinical reasons will be asked to participate in various study tasks with the recording of intracranial EEG (recording of brain waves via electrodes implanted in a participant's brain) during these tasks.
  Interventions: Other: Memory Tasks; Other: Attention/arousal tasks; Other: Language tasks; Other: Visuospatial tasks; Other: Auditory Tasks; Procedure: Brain Stimulation; Other: Social Emotional Task; Other: Recording of facial expressions; Other: Judgement/Impulsivity Task
- Scalp EEG (electrodes are placed on a participant's scalp) (Experimental): Patients with non-invasive scalp electrodes who are admitted to the hospital for clinical reasons will be asked to participate in various study tasks with the recording of their EEG (recording of brain waves via electrodes attached to a participant's scalp) during these tasks.
  Interventions: Other: Memory Tasks; Other: Attention/arousal tasks; Other: Language tasks; Other: Visuospatial tasks; Other: Auditory Tasks; Other: Social Emotional Task; Other: Recording of facial expressions; Other: Judgement/Impulsivity Task
- Normal Controls (Active Comparator): Normal controls will be recruited from family members of patients, from advertisements, or from online tools. There will be no EEG recordings obtained from these participants.
  Interventions: Other: Memory Tasks; Other: Attention/arousal tasks; Other: Language tasks; Other: Visuospatial tasks; Other: Social Emotional Task; Other: Recording of facial expressions; Other: Judgement/Impulsivity Task
- Online Controls (Active Comparator): Certain control subjects will be recruited through Amazon Mechanical Turk. These participants will be given their task on the online platform using Qualtric survey function. The task design will be identical to normal controls who are recruited in-person, with the exception of identifiers. There will be no EEG recordings obtained from these participants.
  Interventions: Other: Memory Tasks; Other: Attention/arousal tasks; Other: Language tasks; Other: Visuospatial tasks; Other: Social Emotional Task; Other: Recording of facial expressions; Other: Judgement/Impulsivity Task

INTERVENTIONS:
Other: Memory Tasks — Participants will be asked to view pictures and videos presented on a computer screen and will be asked to recall the details of presented pictures or videos sometime later.
Other: Attention/arousal tasks — Participants will be asked to perform a continuous performance task, such as continuous addition of numbers. Additionally, participants may be presented with images and may be asked to rate the significance or arousal values for each image.
Other: Language tasks — Participants will be asked to view pictures of actions or things and will be asked to name them. Participants may also be asked to read words or passages.
Other: Visuospatial tasks — Participants will be asked to copy 3 dimensional designs or make judgements of angle size.
Other: Auditory Tasks — Participants will be presented with short, approximately 8-minute clips of music from various genres ( i.e. classical, country, rock, etc.) with an attention task (modified sustained attention to response task) nested within each trial. Participants will receive approximately 8 music stimuli and 1 control stimulus (pink noise) twice over the course of two testing sessions ( 90 mins each). Additionally, participants will be asked to answer questions about their hearing, music preferences/training, and certain demographic information (age, handedness, and language proficiency).
  Arms: Invasive EEG (electrodes are implanted in a participant's brain); Scalp EEG (electrodes are placed on a participant's scalp)
Procedure: Brain Stimulation — A brain stimulator will be used to understand new functions of the brain. Participants will be presented with pictures on a computer screen and may be asked to tell researchers what is seen or remembered by participants. As pictures are viewed by the participants, the brain stimulator may be activated, which would not be something that would be felt by an individual participant.
  Arms: Invasive EEG (electrodes are implanted in a participant's brain)
Other: Social Emotional Task — Participants will be asked to view presented pictures and videos of people engaged in social interaction. Additionally, participants will be presented with the standardized tasks that are designed to help the researchers with understanding the nature of emotions. Some of these images may be emotionally disturbing. If participants are not comfortable viewing such images, they will be asked to refrain from participation in this study.
Other: Recording of facial expressions — Some participants may be asked permission to record the video of their facial expressions during performance of a research task. Generally, this will include only research tasks investigating brain representation of social/emotional information. Automated analysis of facial expression may be used in certain experiments to provide information on experience of emotional states such as happiness and sadness related to the images being presented.
Other: Judgement/Impulsivity Task — Certain study participants may be enrolled into research tasks designed to activate regions important for judgment and impulse control. These tasks will present participants with choices of varying monetary rewards and ask them to make judgements to measure one's tendency to prefer immediate over delayed rewards.

SUMMARY:
This study will enroll patients with epilepsy who are being evaluated for epilepsy surgery and have electrodes implanted in the brain and/or have electrodes on the scalp. Additionally, this study will recruit normal and online controls (participants who do not have epilepsy). Participants will be asked to participate in 1 to 2 (30-90 minutes) daily sessions designed to test aspects of human cognition such as memory, speech, language, feeling, movement, attention, sound perception, and emotions. Generally, this will involve working on a computer, looking at pictures or watching videos, and answering questions. Additionally, participants may be asked to be hooked up to additional equipment such as eye tracker, electrical stimulator, heart rate monitor, sweat monitor or other non-invasive equipment. The overall aim of this study is to use human intracranial electrophysiology (the recording of the electrical activity of the human brain) to study localization and function of the human brain.

DETAILED DESCRIPTION:
This project aims to study the mechanisms of brain function by using Human Intracranial Electrophysiology (HIE) methods and is a continuation of the "Localization of Human Brain Function" study done at Dartmouth-Hitchcock Medical Center (DHMC). HIE refers to the recording of brain signals using electrodes which are surgically inserted into the human brain for the clinical purpose of localizing the origins of epileptic seizures.

Secondary to clinical goals, such patients with intracranial EEG electrodes can be safely recruited to participate in research studies, i.e. the research "piggybacks" on procedures that are performed strictly for a clinical purpose. Brain signals obtained using HIE methods during performance of specific tasks have unique properties rich with insight into the inner workings of the human brain. HIE methods can be used together with electrical brain stimulation (EBS) techniques to better understand relationship between brain and behavior. Furthermore, HIE methods can be recorded together with other non-invasive bio-physiological data streams such as pupillometry, electrodermal activity (EDA), cardiac monitoring, and respiratory monitoring to understand the relationship between the brain and many aspects of human physiology.

ELIGIBILITY:
Patients with Intracranial EEG: Inclusion Criteria

* Patients must be age 18 years or older. There is no upper age limit.
* Patients must have a diagnosis of refractory epilepsy undergoing intracranial EEG recording for clinical purposes.

Patients with Intracranial EEG: Exclusion Criteria

* Patient has additional neurological condition (such as stroke or dementia) or a psychiatric condition (such as active psychosis or suicidal ideation) and are deemed inappropriate for the study
* Patients are not able to provide informed consent for any reason (e.g. encephalopathic, experiencing a seizure)

Patients with Scalp EEG: Inclusion Criteria

* Patients must be age 18 years or older. There is no upper age limit.
* Patients must have a probable diagnosis of epilepsy.

Patients with Scalp EEG: Exclusion Criteria

* Patient has additional neurological condition (such as stroke or dementia) or a psychiatric condition (such as active psychosis or suicidal ideation) and are deemed inappropriate for the study
* Patients are not able to provide informed consent for any reason (e.g. encephalopathic, experiencing a seizure)

Normal Controls: Inclusion Criteria

* Participants must be age 18 years or older. There is no upper age limit.
* Participants must be able to provide informed consent for themselves.

Normal Controls: Exclusion Criteria

• Determined not to be appropriate normal control for the study population

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Using scalp and intracranial EEG, measure changes in electrical activity of the human brain associated with memory. | Evaluated for each patient during monitoring period of approximately 2 weeks.
  Primary objective is to use human intracranial electrophysiology to study localization and function of the human brain. With continuous recording of the electrical activity in participants' brain, study participants will be asked to take part in research tasks involving memory. The researchers will use the information to further the understanding of the exact location of cognitive functions.
Using scalp and intracranial EEG, measure changes in electrical activity of the human brain associated with language. | Evaluated for each patient during monitoring period of approximately 2 weeks.
  Primary objective is to use human intracranial electrophysiology to study localization and function of the human brain. With continuous recording of the electrical activity in participants' brain, study participants will be asked to take part in research tasks involving language. The researchers will use the information to further the understanding of the exact location of cognitive functions.
Using scalp and intracranial EEG, measure changes in electrical activity of the human brain associated with emotions. | Evaluated for each patient during monitoring period of approximately 2 weeks.
  Primary objective is to use human intracranial electrophysiology to study localization and function of the human brain. With continuous recording of the electrical activity in participants' brain, study participants will be asked to take part in research tasks involving emotions. The researchers will use the information to further the understanding of the exact location of cognitive functions.
Using scalp and intracranial EEG, measure changes in electrical activity of the human brain associated with movement. | Evaluated for each patient during monitoring period of approximately 2 weeks.
  Primary objective is to use human intracranial electrophysiology to study localization and function of the human brain. With continuous recording of the electrical activity in participants' brain, study participants will be asked to take part in research tasks involving movement. The researchers will use the information to further the understanding of the exact location of cognitive functions.
Using scalp and intracranial EEG, measure changes in electrical activity of the human brain associated with attention and executive function. | Evaluated for each patient during monitoring period of approximately 2 weeks.
  Primary objective is to use human intracranial electrophysiology to study localization and function of the human brain. With continuous recording of the electrical activity in participants' brain, study participants will be asked to take part in research tasks involving attention and executive function. The researchers will use the information to further the understanding of the exact location of cognitive functions.
Using scalp and intracranial EEG, measure changes in electrical activity of the human brain associated with sound perception. | Evaluated for each patient during monitoring period of approximately 2 weeks.
  Primary objective is to use human intracranial electrophysiology to study localization and function of the human brain. With continuous recording of the electrical activity in participants' brain, study participants will be asked to take part in research tasks involving sound perception. The researchers will use the information to further the understanding of the exact location of cognitive functions.

SECONDARY OUTCOMES:
The degree of correlation between the brain activation and respiratory activity. | Evaluated for each patient during monitoring period of approximately 2 weeks.
  Researchers will investigate the degree of correlation (correlation coefficient or how similar the measurements are) between the human intracranial EEG signals and respiratory activity. The respiratory activity (e.g. breathing rate, oxygen level, etc.) will be measured with non-invasive sensors such as respiratory belt worn around a participant's chest and abdomen as well as a small sensor under their nose.
The degree of correlation between the brain activation and electrodermal activity. | Evaluated for each patient during monitoring period of approximately 2 weeks.
  Researchers will investigate the degree of correlation between the human intracranial EEG signals and electrodermal activity (electrical characteristics of human skin). The electrodermal activity will be measured with non-invasive electrodermal sensors such as wrist or ankle sensors and expressed as a variation in electrical characteristics of participants' skin.
Measure the degree of correlation between the brain activation and sweat variations. | Evaluated for each patient during monitoring period of approximately 2 weeks.
  Researchers will investigate the degree of correlation between the human intracranial EEG signals and sweat volume. The researchers will use use a Q-SWEAT system to noninvasively measure the sweat volume produced during specific study tasks. The Q-SWEAT system has a multicompartmental capsule, which is placed tightly on the skin, often in four standard locations (the dorsal foot, distal leg, proximal leg, and forearm), though any flat, area of skin can be used. Nitrogen gas flows through the inner compartment, and the system detects sweat volume by measuring changes in the relative humidity of returning nitrogen during the recording period.
Measure the degree of correlation between the brain activation and cardiac physiology. | Evaluated for each patient during monitoring period of approximately 2 weeks.
  Researchers will use a CNAP machine (finger sensor) to record heart-rate variability. The CNAP machine will measure the waveform and pressure continuously, which will allow for detection of changes in blood pressure without using an arterial line or other invasive methods. Researchers will investigate the degree of correlation between the human intracranial EEG signals and heart-rate variability, including changes in blood pressure during the performance of study tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof A Bujarski, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No